CLINICAL TRIAL: NCT04334577
Title: Evaluation of the Efficacy of Attenuated Zoster Vaccine, Live From Herpes Zoster in Adults Aged 40 Years or older---a Multicenter, Randomized, Double-blinded,Placebo-controlled Trial Phase III
Brief Title: Study on Efficacy of Attenuated Zoster Vaccine, Live
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: F20190717
Record Dates: First submitted 2020-03-25; First posted 2020-04-06 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attenuated Zoster Vaccine, Live (Experimental): One shot of the vaccine (with live viruses titer >=4.3 LgPFU per dose)
  Interventions: Biological: live attenuated zoster vaccine
- Placebo (Placebo Comparator): one shot of placebo with no live virus
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: live attenuated zoster vaccine — subcutaneous injection
  Arms: Attenuated Zoster Vaccine, Live
Biological: placebo — subcutaneous injection
  Arms: Placebo

SUMMARY:
Varicella-zoster virus (VZV) is a herpesvirus that causes two distinct clinical syndromes. Primary infection is manifested as varicella (chickenpox) , whereas reactivation of latent VZV results in a localized eruption known as herpes zoster. The investigational vaccine of this study is produced by Changchun BCHT biotechnology Co. It's a live attenuated herpes zoster vaccine based on the production process of live attenuated chickenpox vaccine.This study plans to have 25000 adults aged 40 years or older and involves in a randomized, double-blind, placebo-controlled trial . The primary outcome is to evaluate the efficacy of the vaccine against herpes zoster 30 days after vaccination and the safety of the vaccine.

DETAILED DESCRIPTION:
Varicella-zoster virus (VZV) is a herpesvirus that causes two distinct clinical syndromes. Primary infection is manifested as varicella (chickenpox) , whereas reactivation of latent VZV results in a localized eruption known as herpes zoster. The investigational vaccine of this study is produced by Changchun BCHT biotechnology Co. It's a live attenuated herpes zoster vaccine based on the production process of live attenuated chickenpox vaccine.This study plans to have 25000 adults aged 40 years or older and involves in a randomized, double-blind, placebo-controlled trial . The primary outcome is to evaluate the efficacy of the vaccine against herpes zoster 30 days after vaccination and the safety of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* 01 Healthy volunteers aged 40 years or older;
* 02 Able to understand and give informed consent;.
* 03 Able to comply with requirements of all clinical trial protocol for completing the study;
* 04 Axillary temperature ≤37.0 at the time of enrollment;

Exclusion Criteria:

* 05 History of herpes zoster;
* 06 History of vaccination against herpes zoster or varicella ;
* 07 Allergic sensitivity to any of the components (including neomycin) in the study vaccine and a history of severe allergies to other vaccine;
* 08 Premenopausal with positive pregnancy test, pregnant or lactating female, or female planning to become pregnant within 6 months;
* 09 Subjects with congenital history of immunity deficiency (e.g., primary immunoglobulin deficiency, isolated IgA deficiency, etc.) or family history;
* 10 Receipt of immunoglobulins and/or any blood products within the 5 months preceding of study vaccine or planning to receive these products during the study period;
* 11 Immunosuppression resulting from disease,such as immunodeficiency, malignant tumor, HIV infection, organ and bone marrow transplantation, leukemia, lymphoma, Hodgkin's disease caused by low immunity; Receipt of immunosuppressive therapy with corticosteroids (except intermittent topical or inhaled corticosteroids [< 800 g/ d Beclomethasone or equivalent]); Other immunosuppressive/cytotoxic treatments (cancer chemotherapy or organ transplantation);
* 12 Subjects with acute infections (such as mumps, etc.), chronic infections in the acute phase (such as active untreated tuberculosis, etc.) or any advanced immune disease;
* 13 Use of any investigational or non-registered product (drug, biological product or device) other than the study vaccine within 1 month before study vaccination , or planed use during the study period;
* 14 Administration or planned administration of any other immunizations within 1 month before study vaccination or scheduled within the study period after study vaccination.
* 15 Any non-local antiviral active treatment within 1 month prior to vaccination, including but not limited to acyclovir, famciclovir, valacyclovir and ganciclovir;
* 16 Taking certain pharmaceuticals to be like salicylate kind, including aspirin, and diflunisal, or going to take these medicine during the study period.
* 17 history of thrombocytopenia or coagulation disorders that may cause subcutaneous injection contraindications;
* 18 significant diseases or significant underlying diseases (such as pulmonary heart disease, pulmonary edema, hypertension that cannot be effectively controlled with drugs [systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥100 mmHg] that may interfere with or hinder the completion of the study, serious liver and kidney diseases, diabetes with concurrent symptoms, etc.);
* 19 Various infectious, suppurative and allergic skin diseases;
* 20 History of psychiatric and neurological disorders (e.g., depression, epilepsy or convulsion);
* 21 Any other conditions may compromise the safety or availability of participants in the judgment of the investigator.(e.g., malleable psoriasis, chronic pain syndrome, cognitive impairment, severe hearing loss, and other conditions that may interfere with study evaluation).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25000 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-18 (Actual)

PRIMARY OUTCOMES:
The incidence of herpes zoster 30 days to 13 months after vaccination | 30 days - 13 months after the vaccination
  The incidence of herpes zoster diagnosed in participants 30 days to 13 months after vaccination

SECONDARY OUTCOMES:
The incidence of herpes zoster after vaccination | 0 day-13 months after the vaccination
  The incidence of herpes zoster diagnosed in participants after vaccination.
The incidence of laboratory-confirmed herpes zoster 30 days to 13 months after vaccination | 30 days- 13 months after the vaccination
  The incidence of laboratory-confirmed herpes zoster diagnosed in participants 30 days to 13 months after vaccination.
Occurrence of solicited adverse reactions after the vaccination | within 14 days after the vaccination
  Occurrence of solicited adverse reactions within 14 days after the vaccination.
Occurrence of adverse reactions after the vaccination. | within 42 days after the vaccination
  Occurrence of adverse reactions within 42 days after the vaccination.
Occurrence of severe adverse reactions after the vaccination | within 13 months after the vaccination
  Occurrence of severe adverse reactions within 13 months after the vaccination
Geometric mean titre of serum for antibody responses 42 days post-vaccination | 42 days after the vaccination
  Geometric mean titre of Serum for antibody responses at day 42 post-vaccination
Geometric mean fold increase of serum for antibody responses 42 days post-vaccination | 42 days after the vaccination
  Geometric mean fold increase of Serum for antibody responses at day 42 post-vaccination
Four-fold increase rate of serum for antibody responses 42 days post-vaccination | 42 days after the vaccination
  Four-fold increase rate of Serum for antibody responses at 42 day post-vaccination
Geometric mean titre of serum for antibody responses 6 months post-vaccination | 6 months after the vaccination
  Geometric mean titre of Serum for antibody responses at 6 months post-vaccination
Geometric mean fold increase of serum for antibody responses 6 months post-vaccination | 6 months after the vaccination
  Geometric mean fold increase of Serum for antibody responses at 6 months post-vaccination
Four-fold increase rate of serum for antibody responses 6 months post-vaccination | 6 months after the vaccination
  Four-fold increase rate of Serum for antibody responses at 6 months post-vaccination
Geometric mean titre of serum for antibody responses 13 months post-vaccination. | 13 months after the vaccination
  Geometric mean titre of Serum for antibody responses at 13 months post-vaccination
Geometric mean fold increase of serum for antibody responses 13 months post-vaccination. | 13 months after the vaccination
  Geometric mean fold increase of Serum for antibody responses at 13 months post-vaccination
Four-fold increase rate of serum for antibody responses 13 months post-vaccination. | 13 months after the vaccination
  Four-fold increase rate of Serum for antibody responses at 13 months post-vaccination

OTHER OUTCOMES:
The incidence of postherpetic neuralgia （PHN）30 days to 13 months after vaccination | 30 days -13 months after the vaccination
  The incidence of postherpetic neuralgia （PHN）diagnosed 30 days to 13 months after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Master, Principal Investigator — LocationJiangsu Province Center for Disease Control and Prevention; Zhiping Chen, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Jiangsu Province Center for Disease Control and Prevention, Nanjing, Jiangsu
  - Zhejiang Provincial Center for Disease Control and Prevention, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954